CLINICAL TRIAL: NCT01247090
Title: Pilot Study of the Effect of Intradialytic Vasopressin Infusion on Chronic Blood Pressure Control in Hypertensive Patients With End Stage Renal Disease: A Program to Develop a Decisive, Randomized Controlled Trial
Brief Title: Study of the Effect of Intradialytic Vasopressin on Chronic Hypertension in Patients With End Stage Renal Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAE0454 - pilot
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2011-04-28 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Hypertension; End Stage Renal Disease
Keywords: hypertension; end stage renal disease; vasopressin; Arginine Vasopressin; AVP; Pitressin®
MeSH Terms: conditions — Hypertension; Kidney Failure, Chronic; Diabetes Insipidus | interventions — Vasopressins; Arginine Vasopressin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Vasopressin - Very Low Dose (Active Comparator): 0.15 mU per kg per minute
  Interventions: Drug: Vasopressin - Very Low Dose
- Group 2: Vasopressin - Low Dose (Active Comparator): 0.30 mU per kg per minute
  Interventions: Drug: Vasopressin - Low Dose
- Group 3: Placebo (Placebo Comparator): No Dose
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Vasopressin - Very Low Dose — Intradialytic vasopressin (AVP) infusion. The dose is calculated based upon the individual's weight in kilograms. A kilogram is equal to 2.2 pounds. For example, a person who weighs 70 kg (or 154 pounds) would receive a dose equal to 0.15 mU * 70 kg, or 10.5 mU of AVP per minute by infusion at their thrice-weekly dialysis treatments.
  Other Names: Vasopressin Injection; USP (8-L arginine vasopressin); AVP; Pitressin®
  Arms: Group 1: Vasopressin - Very Low Dose
Drug: Vasopressin - Low Dose — Intradialytic vasopressin (AVP) infusion. The dose is calculated based upon the individual's weight in kilograms. A kilogram is equal to 2.2 pounds. For example, a person who weighs 70 kg (or 154 pounds) would receive a dose equal to 0.30 mU * 70 kg, or 21 mU of AVP per minute by infusion at their thrice-weekly dialysis treatments.
  Other Names: Vasopressin Injection; USP (8-L arginine vasopressin); AVP; Pitressin®
  Arms: Group 2: Vasopressin - Low Dose
Drug: Placebo Comparator — Participants in Group 3 will receive an equal volume of normal saline (placebo) infusion during their standard thrice-weekly dialysis treatments.
  Other Names: Normal saline
  Arms: Group 3: Placebo

SUMMARY:
The death rate of patients with endstage renal disease (ESRD) on dialysis each year is 20%, with diseases related to the heart and blood vessels causing about half. About 60% of patients on hemodialysis have high blood pressure, which is poorly controlled in most. Normal blood pressure in these patients greatly improves the chance of living. Increased fluid in the body and bloodstream is a major cause of hypertension in patients with ESRD. Fluid removal during hemodialysis is often limited by symptoms of low blood pressure during the procedure. Therefore the increase in fluid and related high blood pressure is ongoing for many of these patients. Arginine vasopressin (AVP) is a hormone naturally produced by the body which has little effect on blood pressure in healthy people, but acts as a powerful vasoconstrictor (narrows the blood vessels) when blood pressure is threatened. Recent studies have shown when there is too little AVP, patients are more likely to have low blood pressure during dialysis that limits fluid removal, an effect that can be reversed by giving these patients low doses of AVP. This phase II trial will find out which of two doses of AVP (.15 or .30 mU kg-1 min-1), in combination with standard therapy, works best to change interdialytic 44-hour ambulatory systolic blood pressure after 2 weeks. Patients who enroll in this study will be divided into three groups. One group will be given a 0.15 mU kg-1 min-1 dose of AVP at each dialysis session over a 2-week period; the second group will be given AVP 0.3 mU kg-1 min-1 at the same interval; and a third group will be given normal saline (placebo) at the same interval. All patients will be closely monitored for side-effects.

DETAILED DESCRIPTION:
This pilot study originally enrolled a group of 12 subjects (4 subjects per arm) in order to demonstrate feasibility with the primary outcome measure, interdialytic 44-hour ambulatory systolic blood pressure. Data on the original subjects is complete and results are posted.

The data from this study will be used to design and conduct additional study enrollment/extension (24 subjects) in order to make some initial statistical comparisons between groups, which will help establish greater confidence in our novel method for controlling blood pressure in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* End Stage Renal Disease on Hemodialysis greater than 3 months
* Hypertension (Predialysis systolic blood pressure (SBP) greater than 140 mmHg, averaged over preceding 6 dialysis treatments)
* Stable dry weight over preceding 6 dialysis treatments

Exclusion Criteria:

* Age less than 18 years
* Clinically significant vascular disease*
* Predialysis systolic blood pressure (SBP) greater than 200 mmHg or diastolic blood pressure (BP) >110
* Pregnancy
* Long QTc syndrome (an electrocardiogram (ECG) will be performed if unavailable within the last 3 months)

Clinically significant vascular disease is defined as any of the following occurring in the preceding three months: angina, claudication, transient ischemic attack, myocardial infarction, cerebrovascular accident, or decompensated heart failure. Furthermore, patients will be excluded if they have any history of ischemic colitis or Raynaud's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Ganda, M.D., M.S., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Very Low Dose: Very Low Dose: Active Comparator 0.15 mU per kg per minute
- Low Dose: Low Dose: Active Comparator 0.30 mU per kg per minute
- Placebo: No Dose - Placebo Comparator
Period: Overall Study
Arm/Group | Very Low Dose | Low Dose | Placebo
Started | 4 | 4 | 4
Completed | 3 | 3 | 4
Not Completed | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low Dose | Low Dose | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 2
  >=65 years | 4 | 3 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (8.04) | 71.0 (8.98) | 72.3 (8.66) | 73 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 6
  Male | 1 | 1 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 7
  Not Hispanic or Latino | 1 | 3 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 0 | 0 | 2 | 2
  More than one race | 4 | 1 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Interdialytic 44-hour Ambulatory Systolic Blood Pressure Over a 2 Week Follow-up Period
Description: This is designed to measure if the administration of intradialytic AVP will result in change in systolic blood pressure.
Time Frame: Baseline and Two Weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Very Low Dose | Low Dose | Placebo
Number analyzed (Participants) | 4 | 4 | 4
mm Hg | -1.5 (8.6) | -3.7 (27.0) | -0.4 (11.8)

ADVERSE EVENTS:
Time Frame: Two weeks.
Description: Method of systematic assessment: Physician assessment.
Arm/Group | Very Low Dose | Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT01247090/Prot_SAP_000.pdf